CLINICAL TRIAL: NCT00627016
Title: A Phase 3 Multicenter, Randomized, Double-Blind, Parallel Group, Placebo Controlled Trial to Evaluate the Efficacy of TAK-390MR (30 mg QD) Compared to Placebo on Relief of Nocturnal Heartburn in Subjects With Symptomatic Gastroesophageal Reflux Disease (GERD)
Brief Title: A Study of Dexlansoprazole Modified Release Formulation to Treat Night Heartburn
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sr. VP Clinical Sciences, Takeda Global Research & Development Center, Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: T-GD07-170; U1111-1113-9537 (Registry Identifier: WHO)
Record Dates: First submitted 2008-02-21; First posted 2008-02-29 (Estimated); Results first posted 2010-05-06 (Estimated); Last update posted 2011-04-28 (Estimated); Status verified 2011-04

CONDITIONS: Gastroesophageal Reflux
Keywords: Non-Erosive Gastroesophageal Reflux Disease; GERD; heartburn; sleep disturbance; nocturnal Reflux
MeSH Terms: conditions — Gastroesophageal Reflux; Heartburn; Parasomnias | interventions — Dexlansoprazole; Lansoprazole

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexlansoprazole 30 mg QD (Experimental)
  Interventions: Drug: Dexlansoprazole
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexlansoprazole — 30 mg capsule, orally, once daily for 4 weeks
  Other Names: TAK-390; T-168390; TAK-390MR; Kapidex; Dexilant
  Arms: Dexlansoprazole 30 mg QD
Drug: Placebo — 1 capsule, orally, once daily for 4 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether Dexlansoprazole once daily (QD) is effective in treating patients with night heartburn.

DETAILED DESCRIPTION:
This 4 week study of Dexlansoprazole (TAK-390MR) will be conducted by approximately 50 investigators in the United States in patients suffering from night heartburn.

ELIGIBILITY:
Inclusion Criteria:

* Females of childbearing potential who are sexually active must agree to use adequate contraception, and can neither be pregnant nor lactating from Screening throughout the duration of the study.
* History of nocturnal heartburn and GERD associated sleep disturbances prior to screening.
* Meets both of the following criteria: 1) nocturnal heartburn severity of moderate, severe, or very severe on at least 3 of 7 nights and; 2) GERD related sleep disturbances on at least 3 of 7 nights.
* Subjects must have history of symptomatic GERD prior to screening with GERD symptoms that were responsive to acid-suppressive therapy.

Exclusion Criteria:

* Erosive esophagitis visualized during the screening endoscopy.
* Allergy to any proton pump inhibitor drug (lansoprazole, omeprazole, rabeprazole, pantoprazole, esomeprazole), any component of Dexlansoprazole, or Gelusil/antacid.
* Active gastric or duodenal ulcers within 30 days prior to randomization.
* Upper gastrointestinal bleeding within 6 months prior to randomization.
* Co-existing diseases affecting the esophagus (eg, eosinophilic esophagitis, esophageal varices, scleroderma, viral or fungal infection, and/or Barrett's esophagus).
* History of radiation therapy or cryotherapy to the esophagus, caustic or physiochemical trauma such as sclerotherapy to the esophagus.
* Subject requiring dilation for esophageal strictures and/or strictures preventing passage of the endoscope during the screening endoscopy. Schatzki's ring (a ring of mucosal tissue near the lower esophageal sphincter) is acceptable.
* Has another condition that could be the primary cause of the subject's sleep disturbance.
* Evidence of uncontrolled, clinically significant neurologic, cardiovascular, pulmonary, hepatic, renal, metabolic, gastrointestinal, or endocrine disease or other abnormality (other than the disease being studied) which may impact the ability of the subject to participate or potentially confound the trial results.
* Diagnosis of cancer (except basal cell carcinoma) within 5 years of screening.
* Has a condition likely to require surgery during the study.
* Currently diagnosed with acquired immunodeficiency syndrome (AIDS).
* Abnormal clinical laboratory values.
* History of alcoholism or drug addiction.
* Subject who works the night shift.
* Subject who is planning to travel beyond 3 time zones during the study.
* Chronic use (more than 12 doses/month) of non-steroidal anti-inflammatory drugs (NSAIDs), including cyclooxygenase-2 (COX 2) inhibitors within 30 days prior to randomization or anticipated use during the study.
* Use of the following medications during the 14 days prior to randomization or anticipated use during the study: proton pump inhibitors, sucralfate, misoprostol, corticosteroids, prokinetics, anticoagulant therapy, antiseizure medications (other than stable doses), psychotropic medications (other than stable doses), narcotic medications (occasional use allowed), bisphosphonates.
* Use of sleep medications, first generation antihistamines, benzodiazepines, modified cyclic antidepressants, antianxiety medications or drugs with significant anticholinergic effects such as tricyclic antidepressants or drugs with central nervous system effects that could mask perception of symptoms (eg, selective-serotonin reuptake inhibitors, serotonin and norepinephrine reuptake inhibitors). However, subjects who remain on a stable regimen and dose of these medications during the 90 days prior to randomization and who agree to maintain the same regimen and dose during the trial will qualify. Also, short term use of anticholinergics for trial related procedures is not exclusionary. Second generation antihistamines are not excluded.
* Use of histamine (H2) receptor antagonists or antacids (except for trial supplied Gelusil) during the screening period or anticipated use during the treatment period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 305 (Actual)
Dates: Start 2008-03; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Chair — Takeda
Locations (43):
- United States (43):
  - Tucson, Arizona
  - Anaheim, California
  - Garden Grove, California
  - Lancaster, California
  - Oakland, California
  - San Diego, California
  - Sherwood, California
  - Westlake Village, California
  - Jupiter, Florida
  - Miami, Florida
  - New Smyrna Beach, Florida
  - Ocala, Florida
  - St. Petersburg, Florida
  - Zephyrhills, Florida
  - Moline, Illinois
  - Clive, Iowa
  - Wichita, Kansas
  - Metairie, Louisiana
  - Prince Frederick, Maryland
  - Jefferson City, Missouri
  - Egg Harbor Town, New Jersey
  - Great Neck, New York
  - Greensboro, North Carolina
  - Harrisburg, North Carolina
  - Winston-Salem, North Carolina
  - Mogadore, Ohio
  - Oklahoma City, Oklahoma
  - Portland, Oregon
  - Duncansville, Pennsylvania
  - Bristol, Tennessee
  - Chattanooga, Tennessee
  - Johnson City, Tennessee
  - Kingsport, Tennessee
  - Nashville, Tennessee
  - El Paso, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - Odessa, Texas
  - San Antonio, Texas
  - Ogden, Utah
  - Norfolk, Virginia
  - Spokane, Washington
  - Monroe, Wisconsin

REFERENCES:
- [Result] Fass R, Johnson DA, Orr WC, Han C, Mody R, Stern KN, Pilmer BL, Perez MC. The effect of dexlansoprazole MR on nocturnal heartburn and GERD-related sleep disturbances in patients with symptomatic GERD. Am J Gastroenterol. 2011 Mar;106(3):421-31. doi: 10.1038/ajg.2010.458. Epub 2011 Jan 11. PMID 21224838
- See also: Dexilant Package Insert — http://general.takedapharm.com/content/file/pi.pdf?applicationcode=9efb34b3-fb69-4190-a2be-a90b8cb94e25&filetypecode=DEXILANTPI

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at 33 investigative sites in the United States from 07 March 2008 to 20 March 2009.
Pre-assignment Details: Subjects eligible for entry into the Treatment Period were randomized into one of two, once-daily (QD) treatment groups.
Groups:
- Placebo: Placebo capsules, orally, once daily for up to 4 weeks.
- Dexlansoprazole 30 mg QD: Dexlansoprazole 30 mg, capsules, orally, once daily for up to 4 weeks.
Period: Overall Study
Arm/Group | Placebo | Dexlansoprazole 30 mg QD
Started | 153 | 152
Completed | 147 | 146
Not Completed | 6 | 6
Not completed — Adverse Event | 1 | 1
Not completed — Protocol Violation | 0 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Failed Inclusion/Exclusion Criteria | 0 | 1
Not completed — Lack of Efficacy | 1 | 0
Not completed — Placed on Excluded Drugs | 1 | 0
Not completed — Pregnancy | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Dexlansoprazole 30 mg QD | Total
Number analyzed (Participants) | 153 | 152 | 305
Age, Customized [Number; unit: participants]
  <45 years | 75 | 75 | 150
  45 to <65 years | 76 | 75 | 151
  >=65 years | 2 | 2 | 4
Age Continuous [Mean (Standard Deviation); unit: years] | 43.9 (12.45) | 44.6 (11.29) | 44.2 (11.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98 | 97 | 195
  Male | 55 | 55 | 110
Region of Enrollment [Number; unit: participants]
  United States | 153 | 152 | 305
Number of Days with Night Heartburn [Number; unit: participants] — Baseline diary data were summarized using the non-missing diary entries from Study Day -8 to -2, inclusive.
  participants
    0-3 days | 10 | 3 | 13
    4-5 days | 36 | 38 | 74
    6-7 days | 107 | 111 | 218
Number of Nights with Sleep Disturbances Related to Gastroesophageal Reflux Disease (GERD) Symptoms [Number; unit: participants] — Baseline diary data were summarized using the non-missing diary entries from Study Day -8 to -2, inclusive.
  participants
    0-3 Nights | 40 | 33 | 73
    4-5 Nights | 53 | 47 | 100
    6-7 Nights | 60 | 72 | 132

OUTCOME MEASURES:

1. Primary Outcome: Median Percentage of Nights Without Heartburn Over 4 Weeks as Assessed by Daily Diary.
Description: Percentage calculated by the number of heartburn-free nights out of the total number of nights during the treatment period with a diary entry indicating presence or absence of nighttime heartburn in subjects who had ≥1 diary entry indicating presence or absence of nighttime heartburn, as indicated by the subject's daily diary. Subjects indicate the presence (Yes/No) of nocturnal heartburn symptoms in a Daily Electronic Diary. Nights missing diary results were excluded from the numerator and denominator.
Time Frame: 4 Weeks
Population: Analysis was conducted on intent-to-treat subjects (randomized subjects who received at least 1 dose of study drug) who completed at least 1 diary entry for nighttime heartburn during treatment.
Measure: Median (Inter-Quartile Range); unit: Percentage of nights
Arm/Group | Placebo | Dexlansoprazole 30 mg QD
Number analyzed (Participants) | 153 | 151
Percentage of nights | 35.7 (30.0) [7.4 to 61.5] | 73.1 (35.0) [32.0 to 92.3]
Statistical Analysis 1: Comparison: Placebo vs Dexlansoprazole 30 mg QD; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — Statistical significance for the comparison of the primary endpoint was determined at 0.05 level

2. Secondary Outcome: Percent of Subjects With Relief of Night Time Heartburn Over the Last 7 Days of Treatment as Assessed by Daily Diary.
Description: Relief of nighttime heartburn was defined as 6 of 7 nights with no heartburn and at most 1 night with mild heartburn; lack of relief of nighttime heartburn was defined as 2 or more out of 7 nights with heartburn, or 1 night with at least moderate heartburn. Subjects indicate the presence and severity (mild, moderate, severe, or very severe) of nocturnal heartburn in a Daily Electronic Diary. The percentage was calculated as the number of subjects with relief of nighttime heartburn divided by the number of subjects whose relief status could be determined.
Time Frame: Last 7 days of treatment
Population: Analysis was conducted on intent-to-treat subjects (randomized subjects who received at least 1 dose of study drug) who had sufficient diary data to allow for determination of relief status.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Dexlansoprazole 30 mg QD
Number analyzed (Participants) | 148 | 141
Percentage of participants | 19.6 | 47.5
Statistical Analysis 1: Comparison: Placebo vs Dexlansoprazole 30 mg QD; Test type: Superiority or Other; p < 0.001, Fisher Exact — Statistical significance was only declared if the primary endpoint was statistically significant at 0.05 level. The multiplicity between the two secondary endpoints was adjusted by Hommel-Simes method to maintain the overall 0.05 level

3. Secondary Outcome: Percentage of Participants With Relief of Gastro-Esophageal Reflux Disease (GERD) Associated Sleep Disturbances Over the Last 7 Days of Treatment as Assessed by Daily Diary.
Description: Relief of GERD-associated sleep disturbance was defined as 6 of 7 nights with no GERD associated sleep disturbances; lack of relief of GERD-associated sleep disturbance was defined as 2 or more out of 7 nights with GERD-associated sleep disturbance. Subjects indicate the presence (Yes/No) of GERD associated sleep disturbance in a Daily Electronic Diary. The percentage was calculated as the number of subjects with relief of GERD-associated sleep disturbance divided by the number of subjects whose relief status could be determined.
Time Frame: Last 7 days of treatment
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Dexlansoprazole 30 mg QD
Number analyzed (Participants) | 144 | 142
Percentage of participants | 47.9 (29.9) | 69.7 (29.6)
Statistical Analysis 1: Comparison: Placebo vs Dexlansoprazole 30 mg QD; Test type: Superiority or Other; p < 0.001, Fisher Exact — [p-value comment as in outcome 2, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse events summarized were reported after the first dose of study drug and no more than 30 days after the last dose.
Description: Most frequent events are those High Level Terms occurring in at least 5 % of subjects in at least one treatment group.
Arm/Group | Placebo | Dexlansoprazole 30 mg QD
Serious Adverse Events (participants affected / at risk) | 1/153 | 0/152
Other Adverse Events (participants affected / at risk) | 3/153 | 7/152
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=153) | Dexlansoprazole 30 mg QD (N=152)
Abortions Spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=153) | Dexlansoprazole 30 mg QD (N=152)
Upper Respiratory Tract Infections (Infections and infestations) | 3 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication related to study results will be published prior to publication of a multi-center report submitted for publication within 18 months after conclusion or termination of a study at all study sites. Results publications will be submitted to sponsor for review 60 days in advance of publication. Sponsor can require removal of confidential information unrelated to study results. Sponsor can embargo a proposed publication for another 60 days to preserve intellectual property.